CLINICAL TRIAL: NCT04590560
Title: What is the Best Interval to Screen Women 45-49 and 70-74 for Breast Cancer
Brief Title: What is the Best Interval to Screen Women 45-49 and 70-74 for Breast Cancer?
Acronym: MISS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRST174.22
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer, screening, diagnosis, mammography
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: Eligible women signing the written informed consent will be randomized with a 1:1:1 ratio to:
  Arm 1: 1-year screening interval; Arm 2: 2-year screening interval; Arm 3: tailored screening interval on the basis of breast density. Women with very dense breast (BI-RADS category D) will be referred to 1-year interval whereas women with less dense breast to 2-year interval (BI-RADS category A, B, C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1-year screening interval (No Intervention): Women will follow the normal screening program (they will be invited to screen every year)
- 2-year screening interval (Experimental): Women will be invited to screen every two years
  Interventions: Diagnostic Test: screening for breast cancer with tomosynthesis and synthetic 2D mammography performed at different interval compared to actual clinical practice
- 3-tailored screening interval (Experimental): the screening interval will be decided on the basis of breast density. Women with very dense breast (BI-RADS category D) will be referred to 1-year interval whereas women with less dense breast to 2-year interval (BI-RADS category A, B, C)
  Interventions: Diagnostic Test: screening for breast cancer with tomosynthesis and synthetic 2D mammography performed at different interval compared to actual clinical practice

INTERVENTIONS:
Diagnostic Test: screening for breast cancer with tomosynthesis and synthetic 2D mammography performed at different interval compared to actual clinical practice — women will be screened for breast cancer using tomosynthesis and synthetic 2D mammography with an interval defined according to their randomization arm for a follow-up period of 6 years;
  Arms: 2-year screening interval; 3-tailored screening interval

SUMMARY:
Italian, multicenter, study aimed at defining the best interval for screening women 45-49 and 70-74 years for Breast Cancer (BC). This research project includes (1) a controlled, prospective randomized non-inferiority trial to determine the optimal screening interval for women aged 45-49, with and without high mammographic density, (2) a retrospective data collection, with the same purpose, on screening performed by women aged 70-74, and (3) a qualitative research to define the best communication strategy.

DETAILED DESCRIPTION:
According to the 2006 European guidelines, the target age for mammography screening is 50-69 years. For women aged 40-49, effectiveness is less and less certain. For those over 70, the most important concern is overdiagnosis. In Europe, so far, both age groups have been invited to screen only in a few countries and regional areas, including some Italian regions. Recently, new European guidelines have been published, developed in the framework of the European Commission Initiative on Breast Cancer. Although with caution, they recommend screening for both women aged 45-49 and those aged 70-74. The recommended interval is 2 or 3 years in the first case and 3 years in the second. The quality of the evidence on which these recommendations are based is defined as very low. Particularly for women aged 45-49, the new European guidelines indicate the need for a research effort, based on comparative studies, on the effectiveness of different screening intervals. This responsibility also falls on Italy, which is the only European country where women aged 45-49 are invited on an annual basis. Therefore, a research project is proposed which includes (1) a controlled, prospective randomized non-inferiority trial to determine the optimal screening interval for women aged 45-49, with and without high mammographic density, (2) a retrospective data collection, with the same purpose, on screening performed by women aged 70-74, and (3) a qualitative research to define the best communication strategy.

To define the best interval for screening women 45-49 years old a three-arm multicenter randomized non-inferiority trial will be conducted. Women signing the written informed consent will be randomized with a 1:1:1 ratio to:

Arm 1: 1-year screening interval; Arm 2: 2-year screening interval; Arm 3: tailored screening interval on the basis of breast density. Women with very dense breast (Breast Imaging-Reporting and Data System -BI-RADS- category D) will be referred to 1-year interval whereas women with less dense breast to 2-year interval (Breast Imaging-Reporting and Data System -BI-RADS- category A, B, C).

Enrollment will last 2.5 years and all women will be followed for 6 years. 60,000 women will be enrolled.

The primary objective is to compare the cumulative incidence of stage 2 or higher breast cancer between different screening intervals and this will be evaluated at the end of the 6-year follow-up period.

At the same time, data from all women registered in screening archives who have had a negative mammogram at the age of 69-71 years will be collected and analyzed. The data will be retrieved up to the age of 78 and will concern screening mammograms as well as other screening procedures (e.g. biopsies) and also mammograms performed outside the program. Data from screening and outpatient information systems as well as from cancer registries will be used.

To identify the best strategy to communicate changes in screening protocols, especially when the new protocol would be less intensive than the actual one, a qualitative research will be conducted. In particular the following steps will be considered:

* Focus groups for discussing, with women from target population and health care professionals, key arguments identified in a preliminary research (i.e. scientific literature and case-studies research), with particular focus on how they should be translated into communication strategies.
* Pre-test of the study's communication material through web-based semi-structured interviews to eligible women and key-informants.
* Assessment of the effectiveness of the communication material through web-based semi-structured interviews to participants, that may bring insights on how planning communication strategies for the implementation of new screening protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Women invited for their first or second mammography (45 or 46 y/o) presenting for screening;
2. Willingness and ability to comply with scheduled visits;
3. Written informed consent obtained prior to performing any protocol-related procedures.

Exclusion Criteria:

1. Pregnancy status;
2. Personal history of prior breast carcinoma, either invasive or ductal carcinoma in situ (DCIS) diagnosis;
3. Ascertained heredo-familial risk according to the standard family history used in screening programs;
4. Participation in another clinical trial on BC screening;
5. Inability to provide signed informed consent.

Ages: 45 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60000 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To compare the cumulative incidence of stage 2 or higher breast cancer between different screening intervals | 6 years
  Cumulative breast cancer risk will computed as the ratio between the number of stage 2 or higher cancers and the total number of women in the arm. The comparison between arms will be performed using the two proportion Z-test. 95% confidence intervals will also be computed

SECONDARY OUTCOMES:
Participation in screening | 6 years
  number of participating women within 3 months since invitation)/(total invited women). It will be computed for each screening round and overall as average of round participation
contamination proportion (use of mammography) within two screening rounds (in women referred to 2-year interval) | 6 years
  number of women referred to 2-year interval and performing a mammogram within two screening round)/number of women referred to 2-year interval The indicator will be computed only for women randomized to arm 2 and for women referred to 2-year arm in arm 3
Breast cancer detection | 6 years
  number of women with BC diagnosis at screening / number of total screened women
overall recall rate | 6 years
  number of women recalled for further assessment/ number of total screened women.
rate of recall with an invasive procedure (biopsy) | 6 years
  number of women recalled for further assessment with a biopsy/ number of total screened women
interval Breast Cancer rate | 6 years
  number of cancers occurring after a negative mammography and before the date of the next planned appointment/ number of total screened women
cumulative Breast Cancer incidence | 6 years
  Cumulative incidence of BC including baseline test
resource expenditure | 6 years
  Mean costs for each attending woman in every of the following processes:
  Coordination and organization; Invitation; First level mammography; Diagnostic assessment (invasive and non invasive)
prevalence of dense breast in the target population | 6 years
  women with BI-RADS A, B, C, and D/total women included in the tailored arm

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Falcini, MD, Study Chair — IRST IRCCS; Livia Giordano, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza; Marco Zappa, MD, Principal Investigator — ISPRO Firenze
Locations (4):
- Italy (4):
  - Irst Irccs, Meldola (FC), FC
  - Istituto per lo studio, la prevenzione e la rete oncologica (ISPRO), Florence
  - AUSL Romagna, Forlì
  - AOU Città della Salute e della Scienza, Torino

IPD SHARING:
Plan to Share IPD: No